CLINICAL TRIAL: NCT04923581
Title: Effect of Optimized Behavioural Intervention Using The Multi-Phase Optimization Strategy (MOST) on Oral Hygiene Habits of Pre-school Children in Egypt.
Brief Title: Effect of Optimized Behavioural Intervention Using The Multi-Phase Optimization Strategy (MOST).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merna Ihab (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Merna Ihab, Teaching Assistant, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: MOST2021
Record Dates: First submitted 2021-06-08; First posted 2021-06-11 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Dental Caries in Children; Early Childhood Caries
Keywords: MOST, behavioural intervention, early childhood caries

STUDY DESIGN:
Intervention Model Description: A factorial trial following the Multiphase optimization Strategy (MOST)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Condition 1 (Experimental): Participants will receive the constant component only.
  Interventions: Behavioral: Oral Health Behavioral Interventions
- Condition 2 (Experimental): Participants will receive the constant component and storytelling videos .
  Interventions: Behavioral: Oral Health Behavioral Interventions
- Condition 3 (Experimental): Participants will receive the constant component and oral health promotion messages.
  Interventions: Behavioral: Oral Health Behavioral Interventions
- Condition 4 (Experimental): Participants will receive the constant component, oral health promotion messages, and storytelling videos.
  Interventions: Behavioral: Oral Health Behavioral Interventions
- Condition 5 (Experimental): Participants will receive the constant component and motivational interview session.
  Interventions: Behavioral: Oral Health Behavioral Interventions
- Condition 6 (Experimental): Participants will receive the constant component, motivational interview session, and storytelling videos.
  Interventions: Behavioral: Oral Health Behavioral Interventions
- Condition 7 (Experimental): Participants will receive the constant component, motivational interview session, and oral health promotion messages.
  Interventions: Behavioral: Oral Health Behavioral Interventions
- Condition 8 (Experimental): Participants will receive the constant component, motivational interview session, oral health promotion messages and storytelling videos
  Interventions: Behavioral: Oral Health Behavioral Interventions

INTERVENTIONS:
Behavioral: Oral Health Behavioral Interventions — The study will use a factorial design to evaluate the efficacy of three distinct intervention components: Motivational interviewing, storytelling videos and oral health promotion messages, in enhancing mothers' brushing of their preschool children's teeth using fluoridated toothpaste.

SUMMARY:
In the current study, MOST approach is proposed, to engineer an oral health behavior modification intervention, to increase the engagement of mothers in brushing their pre-school children's teeth.

DETAILED DESCRIPTION:
The first phase of this study will be the preparation phase. This will comprise the development of a conceptual framework and conducting a feasibility pilot study consisting of three intervention components: Motivational interviewing (MI), Oral health promotion messages (OHPm), and Storytelling (ST). The second phase of the study is the optimization phase which constitutes a factorial trial of the three selected intervention components (MI, OHPm and ST). Each component will be set at two levels: yes (the intervention is applied) vs no (the intervention is not applied).

ELIGIBILITY:
Inclusion Criteria for mother's of children enrolled in study:

* Has children between 2 and <5 years of age
* Has children with high plaque index scores (PlI≥2 or visible plaque accumulation on maxillary anterior teeth).
* Literate and owns a mobile phone with already set-up or possibility to set-up Whats-App messenger application.
* Willing to participate in the study and receive periodic OHPm and ST videos.

Exclusion Criteria:

* Mothers of children who are not willing to cooperate and show a definite negative behavior (Rating 1 Frankel's classification).
* Mothers of children who are physically disabled or medically compromised.
* Mothers of children in need of emergency dental treatments.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2023-07-08 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change in the plaque index scores of participating children | at baseline, 3 and 6 months
  Measured by the Plaque index of Silness and Loe. Lower plaque scores indicate better oral hygiene
Change in children's frequency of toothbrushing and use of fluoridated toothpaste | at baseline, 3 and 6 months
  Using the World Health Organization questionnaire. Highrr tooth brushing frequency indicates better oral hygiene

CONTACTS AND LOCATIONS:
Overall Officials: Merna Ihab, B.Sc, Principal Investigator — Alexandria University, Faculty of Dentistry; Maha El Tantawi, PhD, Study Director — Alexandria University, Faculty of Dentistry; Wafaa E. El Din, PhD, Study Director — Alexandria University, Faculty of Dentistry
Locations (2):
- Egypt (2):
  - Alexandria University, Faculty of Dentistry, Alexandria
  - Department of Pediatric Dentistry and Dental Public Health, Alexandria University, Faculty of Dentistry, Alexandria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ihab M, El Din WE, Ammar N, Yassin R, El Tantawi M. Using mHealth to promote parents' brushing of preschool children's teeth: a protocol for a randomized factorial trial using the Multi-phase Optimization Strategy (MOST). Trials. 2022 Jan 6;23(1):17. doi: 10.1186/s13063-021-05931-0. PMID 34991701